CLINICAL TRIAL: NCT01555957
Title: Effect of Lipid Intake on Direct Hyperbilirubinemia in Late Preterm and Term Infants With Gastrointestinal Surgical Problems.
Brief Title: Prospective Randomized Clinical Trial of Intravenous Lipids and Cholestasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Rochester (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: URochester
Record Dates: First submitted 2012-03-14; First posted 2012-03-16 (Estimated); Results first posted 2020-12-03 (Actual); Last update posted 2020-12-03 (Actual); Status verified 2020-12

CONDITIONS: Parenteral Nutrition Associated Cholestasis
MeSH Terms: interventions — Fat Emulsions, Intravenous

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: The care taker team provided daily weight to the research pharmacist for calculating the dose of the lipid according to the assignment and then calculated the rate of administration over 18 to 24 hours depending on the volume. The rate and dose was masked to the investigators and participants.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- low dose intravenous lipids (Experimental)
  Interventions: Drug: intravenous lipid
- high dose of intravenous lipids (Placebo Comparator)
  Interventions: Drug: intravenous lipid

INTERVENTIONS:
Drug: intravenous lipid — intravenous given daily for 6 weeks

SUMMARY:
The Investigators hypothesize that increased cumulative amount of lipid intake causes PNAC in late preterm and term neonates with major GI surgical disorders

ELIGIBILITY:
Inclusion Criteria:

All neonates ≥ 34 weeks gestational age with major GI surgical disorders (Gastroschisis, omphalocele, volvulus, trachea-esophageal fistula, duodenal atresia, jejunal atresia, ileal atresia, hirschsprung's disease, anorectal malformation, intestinal obstruction, and GI perforations) requiring surgery admitted to our NICU within first 72 hours will be eligible for this study

Exclusion Criteria:

1. If does not need TPN by 72 hours;
2. Direct hyperbilirubinemia within the first 72 hours after birth;
3. TORCH infections (Toxoplasmosis, CMV, Herpes, Rubella, HIV, etc);
4. Biliary tract disorders leading to direct hyperbilirubinemia;
5. Known metabolic disorders that may be associated with direct hyperbilirubinemia- such as Galactosemia, α-1 antitrypsin deficiency, etc

Max Age: 72 Hours | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2012-02; Primary Completion 2018-10-30 (Actual); Study Completion 2019-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sanjiv Amin, MD, Principal Investigator — University of Rochester; Kunal Gupta, MD, Principal Investigator — University of Rochester
Locations (1):
- University of Rochester, Rochester, New York, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose Intravenous Lipids | High Dose of Intravenous Lipids
Started | 20 | 20
Completed | 20 | 20
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose Intravenous Lipids | High Dose of Intravenous Lipids | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 37.9 (1.1) | 36.7 (1.5) | 37.0 (1.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 13 | 22
  Male | 11 | 7 | 18
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 16 | 15 | 31
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 4 | 5 | 9
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Parenteral Nutrition Associated Cholestasis
Description: Defined as direct bilirubin ≥ 2mg/dl developing within one week of the completion of 6 week randomization period
Time Frame: 7 weeks
Population: Intent to treat analysis
Measure: Count of Participants; unit: Participants
Arm/Group | Low Dose Intravenous Lipids | High Dose of Intravenous Lipids
Number analyzed (Participants) | 20 | 20
Participants | 6 | 6
Statistical Analysis 1: Comparison: Low Dose Intravenous Lipids vs High Dose of Intravenous Lipids; we hypothesized that among ≥ 34 weeks GA infants with GISDs, infants receiving 1g/kg/day S-ILE (lipid minimizing strategy) would have decreased incidence of IFALD compared to those receiving 2g/kg/day S-ILE. We also hypothesized that the rate of rise of DB would be lower among ≥ 34 weeks GA infants with GISDs receiving 1g/kg/day versus 2g/kg/day of S-ILE; Test type: Superiority; p = 0.94, Chi-squared

2. Secondary Outcome: Mean Rate of Change in Direct Bilirubin
Description: Amount of direct (conjugated) bilirubin was measured from sera samples.
Time Frame: baseline, weeks 1, 2, 3, 4, 5 and 6
Measure: Mean (Inter-Quartile Range); unit: mg/dL/week
Arm/Group | Low Dose Intravenous Lipids | High Dose of Intravenous Lipids
Number analyzed (Participants) | 20 | 20
mg/dL/week | 0.16 [0.03 to 0.28] | 0.19 [0.06 to 0.32]
Statistical Analysis 1: Comparison: Low Dose Intravenous Lipids vs High Dose of Intravenous Lipids; We also hypothesized that the rate of rise of direct bilirubin would be lower among ≥ 34 weeks GA infants with GISDs receiving 1g/kg/day versus 2g/kg/day of S-ILE; Test type: Superiority; p = 0.0005, Mixed Models Analysis

ADVERSE EVENTS:
Time Frame: 42 days
Arm/Group | Low Dose Intravenous Lipids | High Dose of Intravenous Lipids
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 0/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Dose Intravenous Lipids (N=20) | High Dose of Intravenous Lipids (N=20)
Cholestasis (Hepatobiliary disorders) | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-01-10): https://cdn.clinicaltrials.gov/large-docs/57/NCT01555957/Prot_SAP_000.pdf
  • Informed Consent Form (2018-01-19): https://cdn.clinicaltrials.gov/large-docs/57/NCT01555957/ICF_001.pdf